CLINICAL TRIAL: NCT03821922
Title: Expression of Endocrine Fibroblast Growth Factor 23 and Hypertensive Disorder Complicating Pregnancy
Brief Title: Fibroblast Growth Factor 23 and Hypertensive Disorder Complicating Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Dongyu Wang, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: FGF23
Record Dates: First submitted 2019-01-23; First posted 2019-01-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: Hypertension, Pregnancy-Induced; FGF23
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnancy-induced pregnancy: Those women (subjects) with pregnancy-induced pregnancy.
- Control: Those healthy pregnant women

SUMMARY:
Hypertensive disorder complicating pregnancy is a set of diseases of pregnancy coexisting with elevated blood pressure. The incidence of it is approximately 5-12%. Pregnancy-induced hypertension is a pregnancy-specific disorder, severely impairing both maternal and fetal health, and the major cause of maternal and perinatal mortality rate increased. But so far, the specific etiology is still unclear.

Recently, fibroblast growth factor 23 (FGF23) has emerged as key endocrine regulators of the metabolism of vitamin D and calcium and phosphorus by combining FGFR-α- Klotho receptor complex. Current studies showed that α- Klotho involved the development of gestational hypertension via the production of endothelial nitric oxide, angiogenesis, and the formation of antioxidant enzymes. On the other hand, vitamin D deficiency during pregnancy has an adverse impact on maternal and fetal health, including gestational hypertension. Therefore, the relationship of the expression of FGF23 and the development of gestational hypertension has attracted the attention of relevant scholars.

The aim of this study is to detect the difference of the expression of FGF23 between the hypertensive women and normal pregnant women.

DETAILED DESCRIPTION:
100 pregnant women with hypertensive disorder complicating pregnancy and 200 normal pregnant control women matched for maternal and gestational age were enrolled in the study. All the subjects underwent antepartum screening in the First Affiliated Hospital of Sun Yat-sen University. Blood samples were obtained after overnight fasting at the first, second and third trimester respectively. Serum FGF23 levels were determined by enzyme-linked immunosorbent assay (ELISA) and were correlated with anthropometric, metabolic, and endocrine parameters.

Data were analyzed by SPSS 20.0 database. The results were expressed as mean ± standard deviations or median with interquartile range. Differences between groups were assessed by Student's unpaired t test, Mann-Whitney U test, or Chi-square test as appropriate. Correlation analysis was performed using the Spearman rank correlation method. To identify independent relationships and adjust the effects of covariates, multiple linear regression analyses were performed. P values of <0.05 were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy;
* Regular antenatal examination from the first trimester;
* Give birth in the university hospital (The 1st affiliated hospital of Sun Yat-sen University)

Exclusion Criteria:

* Younger than 18 years old;
* Older than 40 years old;
* Multiple pregnancy;
* Complicated with other diseases such as hypertension, eclampsia, thyroid diseases, etc.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: university hospital
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression of FGF23 | up to 14 weeks
  expression of FGF23 in different groups in mmol/l
Expression of FGF23 | up to 28 weeks
  expression of FGF23 in different groups in mmol/l
Expression of FGF23 | up to 40 weeks
  expression of FGF23 in different groups in mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Zilian Wang, M.D,PhD, Study Director — O&G Department of the 1st affiliated hospital of Sun Yat-sen University
Locations (1):
- Obstetrics and Gynechology Department of the 1st affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China